CLINICAL TRIAL: NCT05824130
Title: Renal, Metabolic, Hepatic and Bone Outcomes in People Living With HIV and Other Co-morbidities Receiving Different Anti-retroviral Regimens
Brief Title: Clinical Outcomes in HIV With Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grace Lui (Other)
Responsible Party: Sponsor-Investigator, Grace Lui, Honorary Clinical Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: HIV ART study
Record Dates: First submitted 2023-04-05; First posted 2023-04-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- B/F/TAF group: B/F/TAF
- other INSTI-based ART regimen: 1-2 NRTI(s) plus an INSTI other than bictegravir
- non-INSTI-based ART regimen: 2 NRTIs plus NNRTI or protease inhibitor

SUMMARY:
Multi-arm, non-randomized, quality of life

DETAILED DESCRIPTION:
This is a prospective, longitudinal, observational study, performed at a Co-morbidities clinic for PLWH. PLWH with one or more co-morbidities receiving anti-retroviral therapy (ART) will be analyzed for their prevalence and incidence of developing renal, metabolic, hepatic and bone diseases. All participants will be assessed at baseline and followed up for one year, or until change in ART regimen, whichever earlier.

ELIGIBILITY:
Inclusion Criteria:

1. HIV antibody positive
2. Age above 18 years
3. Diagnosis of one or more co-morbidities, including hypertension, diabetes, dyslipidemia, chronic kidney disease, chronic liver disease, and cardiovascular diseases
4. Receiving ART regimen, which consists of B/F/TAF, or 1-2 NRTI(s), plus another anti-retroviral drug, including INSTI other than bictegravir, NNRTI, or protease inhibitor

Exclusion Criteria:

1. Recent diagnosis of AIDS within 6 months
2. Recent hospitalization for management of acute medical problems within 6 months
3. Receiving ART regimens other than the combinations listed in Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV (PLWH)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Renal diseases | Baseline
  Renal disease is defined as glomerular filtration rate (GFR) <60 mL/min/1.73m2, or presence of albuminuria, defined as urine albumin:creatinine >3 mg/mmol, according to Kidney Disease Improving Global Outcomes (KDIGO) categorization of chronic kidney disease.
  Blood will be taken for creatinine and urine for creatinine and albumin levels.
Dyslipidemia | Baseline
  Dyslipidemia is defined as total cholesterol >5.17 mmol/l, triglyceride >1.7 mmol/l, HDL cholesterol <1.03 mmol/l in men and <1.29 mmol/l in women, or LDL cholesterol >4.1 mmol/l, or a history of taking anti-hyperlipidemic drugs, according to the National Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (ATP III) guidelines.
  Fasting blood sample will be taken to measure total, LDL and HDL cholesterol and triglyceride levels.
Cardiovascular risk | Baseline
  High cardiovascular disease risk is defined as QRISK3 >10%.
  QRISK3 will be calculated from QRISK 3 risk calculator at qrisk.org.
Liver steatosis and fibrosis | Baseline
  Liver steatosis is defined as Controlled Attenuated Parameter (CAP) >248 dB/m and significant fibrosis is defined as liver stiffness >9.0 kPa, as measured by transient elastography.
  Transient elastography will be performed to measure CAP and liver stiffness.
Low bone mineral density | Baseline
  Low bone mineral density is defined as T score <-1.0 in men 50 years and in post-menopausal women at either lumbar spine or femoral neck, and Z score <-2.0 in men younger than 50 years and pre-menopausal women, as measured by dual energy X-ray absorptiometry (DXA).
  DXA scan will be performed to measure bone mineral density at lumbar spine and femoral neck.
Health-related quality of life | Baseline
  any severity of problem in the five dimensions of EQ-5D-5L, EQ-5D-5L index and EQ-VAS
  EuroQol 5 level EQ-5D version will be performed to measure the above parameters.

SECONDARY OUTCOMES:
Incidences of Comorbidities | 12 months or at the time of change of ART regimen
  All the above endpoints will be determined at 1 year follow up or at the time of change of ART regimen

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No